CLINICAL TRIAL: NCT00150657
Title: Phase II Trial of Carboplatin/Gemcitabine Plus Bevacizumab in Advanced Non-Small Cell Lung Cancer
Brief Title: Study of Carboplatin/Gemcitabine Plus Bevacizumab in Advanced Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. John Providence Health System (Other)
Collaborators: Genentech, Inc. (Industry); Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVF3121s
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2005-11-29 (Estimated); Status verified 2005-09

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; Carboplatin; Gemcitabine

INTERVENTIONS:
Drug: bevacizumab
Drug: carboplatin
Drug: gemcitabine

SUMMARY:
* this study is being done to find out if the combination of carboplatin and gemcitabine will be more effective in the the treatment of advanced lung cancer if bevacizumab, an agent that blocks tumor blood vessel formation, is added
* the study will measure the time to progression of patients treated with the combination; we hope to show that the addition of bevacizumab improves the time to progression (increases the amount of time before the disease begins to worsen)
* all patients receive all three drugs; there is no placebo

DETAILED DESCRIPTION:
* Patients with advanced (stage IV, and Stage IIIB with effusion) non-small cell lung cancer with non-squamous histology, good performance status, and adequate organ function are eligible.
* Patients with brain metastases, squamous histology, or hemoptysis are excluded.
* All patients must give informed consent.
* Schema gemcitabine 1250 mg/M2 IV day 1,8 carboplatin AUC 5 IV day 1 bevacizumab 15 mg/kg IV day 1 repeated every 21 days for 6 cycles

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven non-small cell lung cancer, newly diagnosed or recurrent after previous surgery and/or radiation therapy
* Stage IV disease or stage IIIB with a malignant pleural effusion
* measurable or evaluable disease
* Performance status 0 or 1 (ECOG)
* adequate renal, hepatic, and bone marrow function
* adequate recovery from previous surgery or radiotherapy
* informed consent

Exclusion Criteria:

* brain metastases
* squamous (epidermoid) histology
* hemoptysis
* central airway disease
* Pancoast tumors
* previous chemotherapy or biologic therapy for lung cancer
* prior malignancy within the previous 5 years except non-melanoma skin cancer or cervical CIS
* pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 2004-11

PRIMARY OUTCOMES:
time to progression

SECONDARY OUTCOMES:
response rate
median survival
one year survival
two year survival
toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Kraut, MD, Principal Investigator — Providence Cancer Institute
Locations (1):
- Providence Cancer Institute, Southfield, Michigan, United States